CLINICAL TRIAL: NCT03530371
Title: Effectiveness of Intranasal Dexmedetomidine for Sedated Auditory Brainstem Response Testing
Brief Title: Intranasal Dexmedetomidine for Sedated Hearing Testing
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fondation Lenval (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17-HPNCL-02
Record Dates: First submitted 2018-05-04; First posted 2018-05-21 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Auditory Brainstem Response
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dexmedetomidine Hydrochloride (Experimental): sedation of patients to perform auditory test
  Interventions: Drug: Dexmedetomidine Hydrochloride

INTERVENTIONS:
Drug: Dexmedetomidine Hydrochloride — intranasal administration of 2.5µg/kg of dexmedetomidine to fall asleep the patients
  Other Names: sedated auditory brainstem response

SUMMARY:
Auditory brainstem response testing is necessary in children who are not able to be tested by classical audiogram, because of their age or an associated retarded psycho-motor development or behavioral and cognitive troubles.

This test needs a perfect immobility of the child, ideally being asleep. This situation is sometimes impossible to achieve in non-cooperative children.

Currently, in the Pediatric Hospital of Nice, the investigators have to do a general anesthesia to perform quality auditory response tests in this kind of patients.

The alternative to a general anesthesia would be a reliable sedative drug, allowing the performance of this diagnostic exam without the need of a hospitalization.

Dexmedetomidine is a sedative drug with an action on the α2 adrenergic receptors. It causes a rapid sedation, similar to the natural sleep and with minimal secondary effects. The possibility of an intranasal administration, avoids the pain and discomfort of a venous access insertion.

DETAILED DESCRIPTION:
Auditory brainstem response testing is necessary in children who are not able to be tested by classical audiogram, because of their age or an associated retarded psycho-motor development or behavioral and cognitive troubles.

This test needs a perfect immobility of the child, ideally being asleep. This situation is sometimes impossible to achieve in non-cooperative children.

Currently, in the Pediatric Hospital of Nice, the investigators have to do a general anesthesia to perform quality auditory response tests in this kind of patients.

The alternative to a general anesthesia would be a reliable sedative drug, allowing the performance of this diagnostic exam without the need of a hospitalization. An intranasal administration avoids the pain and discomfort of a venous access insertion.

Dexmedetomidine is a sedative drug with an action on the α2 adrenergic receptors. It causes a rapid sedation, similar to the natural sleep and with minimal secondary effects. The treatment will be administrated by intranasal way at a dosage of 2,5µg/ kg in a single administration under continuous cardiorespiratory monitoring for 2 hours..

The objective of this work is to evaluate the effectiveness of intranasal dexmedetomidine in the realization of the auditory brainstem response at the child with a cognitive or behavioral disorder

This study will consist of research involving non-randomized, monocentric prospective interventional for a duration of 30 months. Patients from 1 year of age and under 16 years, in context of suspicion of deafness will be included. In view of active queue of otorhinolaryngology service of Nice University Hospital and taking into account lost sight, the investigators can include 60 patients, to have a representative sample of concerned pediatric population.

The primary endpoint will be the rate of children included in the study who could determine the auditory threshold. The non-determination of this threshold (or the determination by resorting to general anesthesia or sedation of another type) regardless of the cause will be considered a failure.

Despite the lack of specific protocols, the applications of dexmedetomidine in children for many diagnostic procedures have been studied in the past few years.

Any prospective study about the efficacy of dexmedetomidine for auditory brainstem response testing has been yet conducted in children

ELIGIBILITY:
Inclusion Criteria:

* Child aged 1 to 15 years old
* American Society Anesthesiologists (ASA) scale patient 1 or 2
* Need to evaluate the child audition in a context of suspicion of deafness, delay of language, global delay of the development, the risk factors of hearing loss
* Impossibility to realize a hearing test by conventional audiogram or behavioral due to a cognitive or behavioral disorder of the child
* Affiliation to social security scheme
* Signature of the authorization documents of the 2 parents or the representative of the parental authority for the participation of the child in the study

Exclusion Criteria:

* Heart disease or heart rhythm disorder
* Pneumopathy or asthmatic crisis in previous 2 weeks in the examination
* Recent used of digoxine or beta-blocker
* Use of anti-epileptic or psychotropic drugs
* Medical history of sleep apnea
* Receptor alpha2 agonist allergy
* Gastrooesophageal reflux disease
* Upper airway abnormality
* Acute cerebrovascular diseases
* Neurologic disorders ( cranial trauma and after neurosurgical operation)
* Recent cerebral vascular accident
* Moyamoya disease
* General anesthesia planned for another procedure

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2019-05-02 (Actual); Primary Completion 2021-11-16 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
quality of diagnostic | 5 minutes after the realization of auditory test
  measure the rate of children for who the auditory threshold is obtained with drug sedation condition.

SECONDARY OUTCOMES:
tolerance of treatment | from drug administration to 24 hours after administration of drug
  The tolerance will measure by the collection of the following undesirable effects:
  * hypotension, bradycardia: deviation of> 20% (systolic pressure for blood pressure) from the normal values defined for the age of the subject under waking conditions
  * hypertension: deviation of> 20% (systolic pressure for blood pressure) from the normal values defined for the age of the subject in waking conditions
  * decrease in oxygenation: decrease in oxygen saturation <90%
  These effects will determinate by cardiorespiratory monitoring during the examination. A routine home phone call on D1 will collect information about possible unexpected side effects.
time of correct sedation | from 5 minutes after drug administration to 5 minutes before auditory test
  measure of time in minutes between the administration of the drug and the obtaining of a correct sedation (4, 5 or 6 of the score of Ramsey).
time of vigilance recovery | from 5 minutes after auditory test to 5 minutes after the patient wake up (Aldrete score equal to 9)
  measure the time between the end of the examination, (defined by the end of the recording and the disconnection of the electrodes) and the recovery of the vigilance of the child , evaluated by the Aldrete score . A score of 9 or more determines a correct recovery of alertness and the possibility of returning home. The child will be reevaluated every 10 minutes until this score is reached.

CONTACTS AND LOCATIONS:
Overall Officials: Ana GIORDANO, MD, Principal Investigator — Hôpitaux Pédiatriques de Nice CHU-LENVAL
Locations (1):
- Hôpitaux pédiatriques de Nice CHU-Lenval, Nice, France

REFERENCES:
- [Derived] Giordano A, Lehner B, Voicu A, Donzeau D, Joulie A, Froissant L, Fontas E, Bailleux S. Intranasal dexmedetomidine for sedation in ABR testing in children: No pain, big gain! Int J Pediatr Otorhinolaryngol. 2024 Jun;181:111981. doi: 10.1016/j.ijporl.2024.111981. Epub 2024 May 11. PMID 38749259